CLINICAL TRIAL: NCT01891708
Title: VEGFRs Predict Bevacizumab Benefit in Advanced Non Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Li Liu (Other)
Responsible Party: Sponsor-Investigator, Li Liu, Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: XHZL02
Record Dates: First submitted 2013-06-19; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Non Small Cell Lung Cancer; Brain Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Bevacizumab; Radiation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — peripheral blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: bevacizumab, standard chemotherapy and radiation — the dose and application model of the three intervention are not specified by the sponsor who just observe the efficacy of the combination application of the three in non small cell lung cancer patients with brain metastasis once enrolled.
  Other Names: Drug:bevacizumab,also Avastine; Drug:standard chemotherapy recommended by clinical guidlines; Radiation

SUMMARY:
a. VEGFRs may be the biomarker which can predict the effect of bevacizumab in non small cell lung cancer

DETAILED DESCRIPTION:
1. non small cell lung cancer (non squamous carcinoma)
2. ECOG 0-1
3. from 18-75 years old

ELIGIBILITY:
Inclusion Criteria:

* non squamous cell non small cell lung cancer
* with measurable disease
* ECOG 0-1

Exclusion Criteria:

- patients received surgery in recent 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced non small cell lung cancer patients with brain metastatic disease
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 months

SECONDARY OUTCOMES:
OS | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Liu, MD, Principal Investigator — Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China